CLINICAL TRIAL: NCT03715777
Title: Electromyographic Study for the Help and Guidance of BoNTA Administration in the Treatment of Chronic Pelvic Floor Pain
Acronym: SEMG
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jose Alberola-Rubio (Other)
Responsible Party: Sponsor-Investigator, Jose Alberola-Rubio, MSc, PhD, Instituto de Investigacion Sanitaria La Fe
Organization: Instituto de Investigacion Sanitaria La Fe (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SEMG
Record Dates: First submitted 2018-10-18; First posted 2018-10-23 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Electromyography; EMG: Myopathy; EMG Syndrome; Pelvic Pain; Pelvic Floor Disorders; Pelvic Pain Syndrome; ElectroPhys: Myopathy
Keywords: BoNTA; Electromyography; EMG; Pelvic Pain; Pelvic Pain Syndrome
MeSH Terms: conditions — Beckwith-Wiedemann Syndrome; Pelvic Pain; Pelvic Floor Disorders | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BoNTA Injection (Experimental): Patients diagnosed with chronic pelvic floor pain, without contraindications for the administration of BoNTA.
  Name of each active substance (INN or proposed INN if available):
  Botulinum toxin type A Clostridium botulinum type A (BoNTA) Pharmaceutical form (use standard terms): Powder and solution for solution for injection Route of administration (relevant to the maximum dose): Intramuscular use Specify total dose : 80 U
  Interventions: Drug: Clostridium botulinum type A (BoNTA)

INTERVENTIONS:
Drug: Clostridium botulinum type A (BoNTA) — Powder and solution for solution for injection Specify total dose: 80 U
  Route of administration:
  Other Names: BoNTA; Clostridium botulinum type A

SUMMARY:
Chronic pelvic pain (CPP) is a common presenting complaint affecting approximately 15-40 % of women aged 18-50 in western countries and 5-43% of women in most developing countries. It is debilitating and has a large socio- economic impact, with a 45%reduction in work productivity, and a 15% increase in absence from work in women with the condition. Botulinum neurotoxin type A (BoNTA) has been suggested to improve pain in muscle spasm, its role in CPP secondary to pelvic floor spasm has gained increasing interest. However, clinicians do not have a diagnosis tool to evaluate the CPP and the BoNTA treatment results.

Design and develop an efficient and simple tool for the diagnosis and detection of pelvic floor muscle (PFM) dysfunction based on superficial electromyography (EMG) and perform 25 EMG registrations sessions in healthy patients and 25 EMG sessions in patients diagnoses with PFM that will be treated with BoNTA to and study the EMG signal before and after BoNTA administration.

ELIGIBILITY:
Inclusion Criteria:

I. Chronic pelvic floor pain (CPD) is defined as pain lasting longer than six months, with absence of proven organic cause and finding of component myofascial present that has been refractory to conventional medical treatment (NSAIDs) II. Sign Informed Consent for the administration of BoNTA III. Authorize to participate in the study IV. Patients who agree not to become pregnant during the duration of the study, using effective contraceptive methods

Exclusion Criteria:

I. Minor II. Pelvic active infection III. General or pelvic malignant disease IV. Psychiatric disease V. Contraindication for the administration of BoNTA VI. Patients who participate in another clinical trial and have been administered a investigational medication within 30 days prior to the planned start of the treatment.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2020-04-29 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale for Pain (VAS) | Week 0 - 12 - 24
  The visual analogue scale or visual analog scale (VAS) is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points.

SECONDARY OUTCOMES:
SF-12 | Week 0 - 12 - 24
  Although Short Form (SF)-12 × 2® has been extensively studied and used as a valid measure of health-related quality of life in a variety of population groups, no systematic studies have described the reliability of the measure in patients with behavioral conditions or serious mental illness (SMI).
Index of Female Sexual Function (IFSF) | Week 0 - 12 - 24
  The Index of Female Sexual Function (IFSF) is a brief questionnaire measure of sexual functioning in women. It was developed for the specific purpose of assessing domains of sexual functioning (e.g. sexual arousal, orgasm, satisfaction, pain) in clinical trials.
The Patient Global Impression of Improvement (PGI-I) | Week 0 - 12 - 24
  The Patient Global Impression of Improvement (PGI-I) is a global index that may be used to rate the response of a condition to a therapy (transition scale). It is a simple, direct, easy to use scale that is intuitively understandable to clinicians
The Clinical Global Impressions Scale (CGI-I) | Week 0 - 12 - 24
  The Clinical Global Impressions scale (CGI) consists of three different global measures: Severity of illness: (CGI-S); Global Improvement (CGI-I); Efficacy index The CGI-I score generally tracks with the CGI-S such that improvement in one follows the other; CGI-S and CGI-I scores can occasionally be dissociated
Electromyography of pelvic floor | Week 0 - 12 - 24
  Electromyography (EMG) is an electrodiagnostic medicine technique for evaluating and recording the electrical activity produced by skeletal muscles

CONTACTS AND LOCATIONS:
Overall Officials: Fco Jose FJ Nohales, MD, phD, Principal Investigator — Hospital Universitario La Fe
Locations (1):
- Hosptial Universitario y Politécnico La Fe, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: European Union Clinical Trials Register — https://www.clinicaltrialsregister.eu/ctr-search/trial/2017-000642-22/ES